## FHIR-ed Up for Tobacco Cessation

## NCT06292130

Statistical Analysis Plan: R43HL156588

December 15, 2024

## Statistical Analysis Plan

This study involved a single-group, pre-post design. Paired t-tests were used to determine the effect of the *refresh* intervention on the primary and secondary outcomes. The primary outcome was change, from pretest (baseline) to posttest (30 day follow-up), in psychosocial expectancies for smoking. Secondary outcome measures include change in confidence to quit smoking between pretest (baseline) and posttest (30 day follow-up) assessments. Cohen's d was used to assess the magnitude of the differences.